CLINICAL TRIAL: NCT01526356
Title: Phase II Study of Topical Rapamycin to Erase Angiofibromas in TSC-Multicenter Evaluation of a Novel Therapy
Brief Title: Topical Rapamycin to Erase Angiofibromas in TSC
Acronym: Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mary Kay Koenig, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-11-0501; Department of Defense USAMRMC (Other Grant/Funding Number: W81XWH-11-1-0240)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Angiofibromas; Tuberous Sclerosis
Keywords: Angiofibroma; Tuberous Sclerosis; Rapamycin; Sirolimus; mTOR
MeSH Terms: conditions — Angiofibroma; Tuberous Sclerosis | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Cream only
  Interventions: Drug: Placebo
- 0.1 % Rapamycin (Active Comparator): 0.1% Rapamycin cream
  Interventions: Drug: Rapamycin
- 1% Rapamycin (Active Comparator): 1% Rapamycin cream
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Placebo — Study cream is applied nightly to the affected areas on the face.
  Other Names: Rapamycin
  Arms: Placebo
Drug: Rapamycin — Study cream is applied nightly to the affected areas on the face. Low Dose
  Arms: 0.1 % Rapamycin
Drug: Rapamycin — Study cream is applied nightly to the affected areas on the face. High Dose
  Arms: 1% Rapamycin

SUMMARY:
The study is a multi-center prospective, randomized, double-blind, placebo-controlled evaluation of the safety and efficacy of a topically applied formulation of rapamycin to cutaneous angiofibromas in subjects with Tuberous Sclerosis Complex (TSC). Subjects will apply either the topical vehicle containing rapamycin or the topical vehicle alone nightly to their angiofibromas for six months.

The primary goal of this study is to evaluate the efficacy of the topical medication for reduction of cutaneous angiofibromas in patients with TSC. The secondary goal of this study is to confirm the safety of the topical medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to comply with all trial requirements.
* Subject has a diagnosis of TSC and has visible facial angiofibromas.
* Female subjects of child bearing potential must not be pregnant and must agree to use appropriate contraceptive methods .

Exclusion Criteria:

* Subject is currently receiving therapy with Rapamycin.
* Subject is receiving any form of immunosuppression or has previously experienced immune dysfunction.
* Subject is currently participating in or has participated within the last 30 days in a clinical trial involving an investigational drug.
* Subject has a known hypersensitivity to either the vehicle or Rapamycin.
* Subject is a pregnant or nursing female.
* Subject has other dermatologic conditions that would preclude or prevent adequate assessment of changes to their facial angiofibromas.
* Subject has had laser surgery, cryotherapy, or other dermatologic treatment to their facial angiofibromas within the previous 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Koenig, MD, Principal Investigator — The University of Texas Medical School at Houston; Hope Northrup, MD, Principal Investigator — The University of Texas Medical School at Houston
Locations (10):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Jack & Julia Center for TSC at Oakland Children's Hospital & Research Center, Oakland, California
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Herscot Center for Adults and Children with TSC Massachusetts General Hospital, Boston, Massachusetts
  - Clinic Without Walls, Saint Paul, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Scottish Rite Hospital, Dallas, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
- Sydney Children's Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Koenig MK, Bell CS, Hebert AA, Roberson J, Samuels JA, Slopis JM, Tate P, Northrup H; TREATMENT Trial Collaborators. Efficacy and Safety of Topical Rapamycin in Patients With Facial Angiofibromas Secondary to Tuberous Sclerosis Complex: The TREATMENT Randomized Clinical Trial. JAMA Dermatol. 2018 Jul 1;154(7):773-780. doi: 10.1001/jamadermatol.2018.0464. PMID 29800048

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo
Started | 59 | 63 | 57
Completed | 51 | 53 | 45
Not Completed | 8 | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo | Total
Number analyzed (Participants) | 59 | 63 | 57 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.2 (13.0) | 21.7 (12.4) | 20.3 (14.3) | 20.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 29 | 99
  Male | 23 | 29 | 28 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Facial Angiofibroma Grading Scale (AGS) Score
Description: Subject's lesion/s will be digitally photographed before initial application (visit 1), at each study visit (visits 2 through 6), and immediately prior to study termination (visit 7). Following completion of the study, all photographs will be evaluated by two independent dermatologists blinded to both the treatment arm and the stage of treatment. The dermatologists will assess each photograph's appearance using the facial Angiofibroma Grading Scale (AGS), which assesses the forehead, nose, cheeks, and chin for erythema, average lesion size, lesion density, and percent involvement, as well as presence of any pedunculated angiofibromas. A total score is reported with a range of 0 to 202, with higher scores representing a worse outcome.
Time Frame: baseline, 6 months
Population: This data was not collected for 12 in the 1% rapamycin arm, 17 in the 0.1% rapamycin arm, and 17 in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo
Number analyzed (Participants) | 47 | 46 | 40
score on a scale | -13.89 (20.86) | -12.71 (20.24) | -1.39 (14.64)

2. Secondary Outcome: Photo Readers' Rating (Better, Same, or Worse) of Paired Baseline and End-of-trial (EOT) Photographs for Each Patient
Time Frame: baseline, 6 months
Population: This data was not collected for 4 in the 1% rapamycin arm, 5 in the 0.1% rapamycin arm, and 6 in the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo
Number analyzed (Participants) | 55 | 58 | 51
Participants
  better | 45 | 38 | 13
  same | 5 | 11 | 15
  worse | 5 | 9 | 23

3. Secondary Outcome: Change in Quality of Life (QOL) Questionnaire Scores as Assessed by the Dermatology Life Quality Index (DLQI)
Description: The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above. Each question is scored from 0 to 3, giving a possible total score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Time Frame: baseline, 6 months
Population: This data was not collected for 29 in the 1% rapamycin arm, 34 in the 0.1% rapamycin arm, and 35 in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo
Number analyzed (Participants) | 30 | 29 | 22
score on a scale | -1.5 (4.4) | -3.2 (5.0) | -1.6 (4.5)

4. Secondary Outcome: Change in Quality of Life (QOL) Questionnaire Scores as Assessed by the Children's Dermatology Life Quality Index (CDLQI)
Description: The Children's Dermatology life Quality Index (DLQI) is validated from the age of four years to 16 years. It is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question is scored from 0 to 3, giving a possible total score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Time Frame: baseline, 6 months
Population: This data was not collected for 46 in the 1% rapamycin arm, 57 in the 0.1% rapamycin arm, and 48 in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo
Number analyzed (Participants) | 13 | 6 | 9
score on a scale | -0.2 (4.1) | -1.7 (3.1) | -1.8 (2.6)

5. Secondary Outcome: Change in Quality of Life (QOL) Questionnaire Scores as Assessed by the Family Dermatology Life Quality Index (FDLQI)
Description: The Family Dermatology life Quality Index (FLQI) is designed for adult (more than 16 years of age) family members or partners of patients (of any age) with any skin disease. It is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question is scored from 0 to 3, giving a possible total score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Time Frame: baseline, 6 months
Population: This data was not collected for 41 in the 1% rapamycin arm, 35 in the 0.1% rapamycin arm, and 38 in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo
Number analyzed (Participants) | 18 | 28 | 19
score on a scale | -2.2 (3.2) | -1.8 (5.2) | 0.3 (3.4)

6. Other Pre Specified Outcome: Number of Events of Dermatologic Sensitivity at the Site of Application
Description: Dermatologic sensitivity includes pain, pruritis, or erythema at the application site.
Time Frame: 6 months
Measure: Number; unit: number of events
Arm/Group | Placebo | 0.1 % Rapamycin | 1% Rapamycin
Number analyzed (Participants) | 59 | 63 | 57
number of events
  Application site pain | 6 | 2 | 1
  Application site pruritis | 5 | 0 | 1
  Application site erythema | 2 | 1 | 0

7. Other Pre Specified Outcome: Number of Participants With Systemic Uptake of Topically Applied Rapamycin
Description: Blood levels checked to confirm the lack of systemic rapamycin.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Rapamycin | 0.1 % Rapamycin | Placebo
Number analyzed (Participants) | 59 | 63 | 57
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious adverse events were determined to be unrelated to study drug.
Arm/Group | Placebo | 0.1 % Rapamycin | 1% Rapamycin
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/63 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/63 | 2/57
Other Adverse Events (participants affected / at risk) | 10/59 | 18/63 | 22/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | 0.1 % Rapamycin (N=63) | 1% Rapamycin (N=57)
cholecystectomy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Subependymal Giant Cell Astrocytoma (SEGA) resection (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | 0.1 % Rapamycin (N=63) | 1% Rapamycin (N=57)
Application site pain (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 6 (6)
Application site pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Application site acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Cutaneous eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Application site erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Application site irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Application site papules (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Application site paraesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Mouth ulceration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes